CLINICAL TRIAL: NCT03757624
Title: TISSUE SHRINKAGE DEPENDS ON FORMOL SOLUTION IN DIFFERENT GASTRIC LOCATIONS
Acronym: SHRINKAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANIL ERGIN.
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Shrinking Stomach
Keywords: shrinkage; formol; stomach; gastric wall
MeSH Terms: interventions — els extra low shrinkage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric specimen measurements after 24 hours from % 10 formol (Active Comparator): Gastric specimens of patients who will undergo to Laparoscopic Sleeve Gastrectomy ,will examine after formol solution
  Interventions: Procedure: shrinkage
- Gastric specimen measurements after surgery in operating room (Active Comparator): Gastric specimens of patients who will undergo to Laparoscopic Sleeve Gastrectomy ,will examine after surgery in operating room peroperatively
  Interventions: Procedure: shrinkage

INTERVENTIONS:
Procedure: shrinkage — shrinkage of gastric specimen in %10 formol solution after Laparoscopic Sleeve Gastrectomy

SUMMARY:
Generally % 10 formol solution is use to do fixation to all specimens after the surgical operations for the pathological evaluation. It is known that the formol solution cause amount of shrinkage in the tissue volume . This effect of formol solution had researched in colon,breast and prostate previously. But there is no evidence about stomach. The purpose of this research is that find out the formol effect to the gastric tissue and detect the shrinkage percent.

DETAILED DESCRIPTION:
All gastric specimens which removed after Laparoscopic Sleeve Gastrectomy will open from the major curvature and spread down to the table.in operating room..3 cm x 3 cm three tissue samples will collect from the specific locations. These three locations are ; fundus( 1 cm from the top of staple line) , corpus (middle of the major curvature , antrum ( 1 cm far from the bottom of staple line ). All these points 5 mm far from the major curvature. 6 samples will prepare totally. 2 samples for each location ; one mucosa and one all layer of gastric wall for each location .These 3 points will examine about wall thickness(mucosa- submucosa-muscularis propria -serosa ) After saving the measurements in operating room;the gastric specimen will deliver to a pathologist to put the specimen into the % 10 formol solution. After 24 hours ;pathologist will save all of new measurements same in operating room. The measurements of sample are ;height , length , width . After the completion of the measurements the investigator will compare the results found in operating room in fresh specimen with pathologist 's results after formol. After that the investigator will be able to decide the shrinkage of gastric tissue in % 10 formol solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old who will undergo to Laparoscopic Sleeve Gastrectomy

Exclusion Criteria:

* Patients who has to undergo another bariatric surgery type peroperatively
* Deformation of gastric specimen while removing from the abdomen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
shrinkage in gastric tissue | 24 hours
  shrinkage of gastric specimen in %10 formol solution after Laparoscopic Sleeve Gastrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No